CLINICAL TRIAL: NCT01521104
Title: The Value of NBI in Stratifying Patients for Endoscopic Resection or Surgery
Brief Title: The Value of Narrow Band Imaging in Stratifying Patients for Endoscopic Resection or Surgery
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaobo Li, Shanghai Institute of Digestive Disease，Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Other Study IDs: rjxhnk02
Record Dates: First submitted 2012-01-25; First posted 2012-01-30 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Colorectal Neoplasms
Keywords: narrow band imaging（NBI）; colorectal lesions; predicting histology
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All the lesions will be removed endoscopically or surgically and examined histologically by an independent gastrointestinal pathologist.
  Histological diagnosis is determined according to the World Health Organization (WHO) criteria.Pedunculated lesions are categorized according to Haggitt's classification.
Oversight: Data Monitoring Committee: No

SUMMARY:
Magnification narrow band imaging (NBI) can make accurate evaluation in in predicting of invasive depth of colorectal neoplasia.

DETAILED DESCRIPTION:
NBI could be used in stratifying patients for endoscopic resection or surgery and got an accurate evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with more than one lesion ≧6mm

Exclusion Criteria:

* Patients with chronic inflammatory bowel disease,
* advanced cancer,
* insufficient bowel preparation,
* familial adenomatous polyposis (FAP)
* Lesions ≦ 5mm and submucosal tumor (SMT).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive adult patients undergo colonoscopy and find out more than one lesion ≧ 6mm from Jan 2009 to Dec 2010
Sampling Method: Non-Probability Sample
Enrollment: 565 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)